CLINICAL TRIAL: NCT03567772
Title: Videogame Assisted Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Yusup subagio sutanto, Head of Pulmonary Department, medical faculty of Universitas Sebelas Maret, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USebelasMaret
Record Dates: First submitted 2018-06-11; First posted 2018-06-26 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Video-game assisted rehabilitation; COPD; Exercise tolerance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wiifit Nintendo video game (Experimental): Pulmonary rehabilitation program using video games exercise from Nintendo
  Interventions: Device: Wiifit Nintendo video game; Other: Pulmonary rehabilitation program
- Pulmonary rehabilitation program (Active Comparator): Pulmonary rehabilitation program with ergometer cycle
  Interventions: Other: Pulmonary rehabilitation program

INTERVENTIONS:
Device: Wiifit Nintendo video game
  Arms: Wiifit Nintendo video game
Other: Pulmonary rehabilitation program

SUMMARY:
Pulmonary rehabilitation programs (PRP) are a key factor of comprehensive management of patients with chronic obstructive pulmonary disease (COPD). Interactive game-based systems have been proposed to improve effects and/or compliance to PRP. The aim of this study is to evaluate the effectiveness of wiifit nintendo as a PRP tool in COPD patients with a randomized controlled trial methods. The patients were divided into experimental (EG) and control (CG) group. The EG performed wiifit program (yoga, strength training, aerobic exercise) twice a week for 6 weeks, the CG performed cycle ergometer twice a week for 6 weeks. The investigators evaluated pre and post treatment: Six-minute walking test, Transitional Dyspnea Index, and Saint George Respiratory Questionnaire.The hypothesis are the EG able to show improvement in exercise tolerance, dyspnea, and quality of life.

DETAILED DESCRIPTION:
In this randomised clinical trial (RCT) subjects were assigned to two groups: the Experimental Group (EG) received a hospital based outpatient PRP and Wii Fit videogame program; the Control Group (CG) received only a standard hospital based outpatient PRP. Researchers evaluating results and patients were not blind to treatment. Patients maintained their usual drug medication according to accepted Guidelines.

Patients of both groups received for six weeks three weekly 30-minute sessions of supervised standard cycle exercise training at outpatient clinics under the supervision of doctors and nurses. Oxygen pulse oximetry (SpO2), arterial blood pressure, heart rate (HR) and dyspnoea (by a 10-point modified Borg scale) were monitored.

In addition to each session of exercise training, patients of EG performed also 30 minute session of supervised video-game assisted program in a dedicated room equipped with Wii Nintendo, balance board, and flatscreen television. Participants played 3 different games per session:

1. Yoga with "deep breathing" and "half moon" : patients performed technique of breathing and held a particular pose or series of poses for 10 minutes.
2. "torso twist" : a strength training exercise in which patients perform a number of repetitions of the selected exercise.
3. aerobic exercises "free run": the patient runs in place while keeping the connected Wii Remote in his or her pocket, which acts as a pseudo-pedometer.

The primary outcome measure was the 6MWT. Results are shown as mean (Standard Deviation: SD) for continuous and as numbers (percentage frequency) for discrete variables. To determine the sample size, an earlier study showed a post-program 70.4 (18.3) meter mean increase in 6MWT.

The study hypothesis was therefore to observe a 30 m post-PRP change in both groups. To obtain a 90% study power and an alpha error less than 5%, a minimum sample size of 12 patients completing the study was required in each group.

To obtain this result investigators estimated an allocation sample size of 40 patients, considering a 20% drop out rate.

Unpaired t test, Kruskall-Wallis H test, and X2 analyses for dichotomous variables were used when appropriate for comparison between groups to test any baseline difference.

The two-way repeated measures ANOVA was carried out to compare the improvements of both groups.

Chi-square test was used to compare continuous and categorical variables. A p value less than 0.05 was considered as statistically significant. Analyses were performed using a specific package (SPSS for Windows latest version, Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* COPD based on GOLD guidelines
* COPD stable (no exacerbation in the four weeks prior to study)

Exclusion Criteria:

* refusal to participate
* participation in a PRP during the previous 6 months
* severe concomitant comorbidities such as ischaemic cardiac disease, chronic heart failure, orthopaedic and/or neuromuscular diseases interfering with their ability to walk.

Dropout criteria:

* acute exacerbation
* inability or unwillingness to follow the research program.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2014-03-30 (Actual); Study Completion 2014-07-30 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance | 6 weeks
  Before and after the pulmonary rehabilitation program the exercise tolerance is measured by Six minute walking distance test (6MWT). Participants have to walk as far as possible for 6 minutes. Participants will walk back and forth in the hallway. Six minutes is a long time to walk, participants are permitted to slow down, to stop and to rest as necessary. The scale will be in meter (m). Higher values represent a better outcome

SECONDARY OUTCOMES:
Health related quality of life: St George's Respiratory Questionnaire (SGRQ) | 6 weeks
  Before and after the pulmonary rehabilitation program, health related quality of life is measured by St George's Respiratory Questionnaire (SGRQ). Three component scores are calculated: symptoms; activity; impacts. One total score is also calculated. Each questionnaire response has a unique empirically derrived weight. The lowest possible weight is zero and the highest is 100. Higher values represent a worse outcome
Dyspnea | 6 weeks
  Before and after the pulmonary rehabilitation program the dyspnoea was assessed by means of the Baseline (BDI) and Transitional (TDI) dyspnoea index. Three component scores are calculated: functional impairment; magnitude of task; magnitude of effort. The lowest possible score is -3 and the highest score is +3. Higher values represent a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rima, Dr, Study Director — Pulmonary Department of Medical faculty Universitas Sebelas Maret, Surakarta Indonesia
Locations (1):
- Pulmonary department of medical faculty Universitas Sebelas Maret, Surakarta, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Maltais F, LeBlanc P, Jobin J, Berube C, Bruneau J, Carrier L, Breton MJ, Falardeau G, Belleau R. Intensity of training and physiologic adaptation in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 Feb;155(2):555-61. doi: 10.1164/ajrccm.155.2.9032194.
- [Background] Mahler DA, Weinberg DH, Wells CK, Feinstein AR. The measurement of dyspnea. Contents, interobserver agreement, and physiologic correlates of two new clinical indexes. Chest. 1984 Jun;85(6):751-8. doi: 10.1378/chest.85.6.751. PMID 6723384
- [Background] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Background] Jones PW. Health status measurement in chronic obstructive pulmonary disease. Thorax. 2001 Nov;56(11):880-7. doi: 10.1136/thorax.56.11.880. PMID 11641515
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] de Torres JP, Pinto-Plata V, Ingenito E, Bagley P, Gray A, Berger R, Celli B. Power of outcome measurements to detect clinically significant changes in pulmonary rehabilitation of patients with COPD. Chest. 2002 Apr;121(4):1092-8. doi: 10.1378/chest.121.4.1092. PMID 11948037
- [Background] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Background] Cote CG, Celli BR. Pulmonary rehabilitation and the BODE index in COPD. Eur Respir J. 2005 Oct;26(4):630-6. doi: 10.1183/09031936.05.00045505. PMID 16204593
- [Background] Turnip H, Ratnawati A, Tulaar A, Yunus F, Kekalih A. Comparison of the effects of treadmill and ergocycle exercise on the functional capacity and quality of life of patients with chronic obstructive pulmonary disease. Med J Indonesia. 2014; 23: 42-47
- See also: 2018 Global strategy for prevention, diagnosis and management of COPD. http://goldcopd.org/gold-reports/. Accessed April 26, 2018. — http://goldcopd.org/gold-reports/